CLINICAL TRIAL: NCT02521961
Title: Developing an Intervention to Reduce Stress and Improve Quality of Life in Underserved Urban Latina Breast Cancer Survivors
Brief Title: Support Group Program in Improving Quality of Life in Underserved Urban Latina Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 9425; NCI-2015-01183 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P30CA015704 (NIH)
Record Dates: First submitted 2015-08-06; First posted 2015-08-13 (Estimated); Last update posted 2018-10-05 (Actual); Status verified 2018-10

CONDITIONS: Breast Carcinoma; Cancer Survivor
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (support group sessions) (Experimental): Participants attend support group sessions over 1-1.5 hours once weekly for 10 weeks. The sessions include facilitated discussions among participants about the following topics: stress management and emotional coping strategies, nutrition and physical activity, sexuality and body image, medical advocacy, self-care and social support. Participants receive a binder in which the rationale for each topic, techniques learned, and activities completed during each session will be summarized and are shown a Chair-robics DVD.
  Interventions: Other: Informational Intervention; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Procedure: Support Group Therapy
- Arm II (control) (Active Comparator): Participants receive one phone call to arrange a follow-up with the promotora, a note acknowledging their participation in the study, and a community resource booklet. Participants are then yoked into one of the 3 intervention groups and asked to attend a 30 minute session similar to Arm I.
  Interventions: Other: Informational Intervention; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Informational Intervention — Watch a Chair-robics DVD
  Arms: Arm I (support group sessions)
Other: Informational Intervention — Receive community resource booklet
  Arms: Arm II (control)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Procedure: Support Group Therapy — Attend support group sessions
  Arms: Arm I (support group sessions)

SUMMARY:
This randomized clinical trial studies a support group program in improving quality of life in underserved urban Latina breast cancer survivors. A psychosocial support group program may help reduce distress and improve health-related quality of life in underserved urban Latina breast cancer survivors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the effect of the support program for Latina breast cancer survivors using validated measures of health-related quality of life.

II. Evaluate the effect of the support program for Latina breast cancer survivors using validated measures of general distress.

SECONDARY OBJECTIVES:

I. A brief qualitative assessment will evaluate the perception of the program among intervention participants using a brief survey.

OUTLINE: Participants are randomized to 1 of 2 arms.

ARM I: Participants attend support group sessions over 1-1.5 hours once weekly for 10 weeks. The sessions include facilitated discussions among participants about the following topics: stress management and emotional coping strategies, nutrition and physical activity, sexuality and body image, medical advocacy, self-care and social support. Participants receive a binder in which the rationale for each topic, techniques learned, and activities completed during each session will be summarized and are shown a Chair-robics digital video disc (DVD).

ARM II: Participants receive one phone call to arrange a follow-up with the promotora, a note acknowledging their participation in the study, and a community resource booklet. Participants are then yoked into one of the 3 intervention groups and asked to attend a 30 minute session similar to Arm I.

ELIGIBILITY:
Inclusion Criteria:

* Latino
* Spanish-speaking
* Diagnosed with breast cancer
* A current resident of either King, Snohomish or Pierce counties in Washington State with the intent of remaining a resident for at least 3 months following study enrollment
* Additionally, at time of enrollment, participants must be post-treatment (with the exception of adjuvant therapy) for their primary cancer and not actively undergoing treatment for a secondary, metastatic, or recurrence of cancer (local or distant)
* There will be no restrictions on time since diagnosis for participants

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-02-03 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2017-07-01 (Actual)

PRIMARY OUTCOMES:
Adherence assessed using weekly attendance records | Up to 10 weeks
  Skewed data will be log transformed or other appropriate transformations performed as necessary. Simple associations between demographic variables and outcome variables will be conducted to determine the need for control variables. Significant pre- to post-intervention change in psychosocial outcomes will be analyzed using the repeated measures linear mixed model. All analyses will be two-tailed and held to a significance level of alpha = 0.05. Post-hoc analyses will otherwise be conducted as appropriate pending the outcome of the initial primary analyses.
Change in acculturation to reflect language use and media, as well as ethnic social relationships, assessed using the Short Acculturation Scale for Hispanics | Baseline to up to 10 weeks
  Skewed data will be log transformed or other appropriate transformations performed as necessary. Simple associations between demographic variables and outcome variables will be conducted to determine the need for control variables. Significant pre- to post-intervention change in psychosocial outcomes will be analyzed using the repeated measures linear mixed model. All analyses will be two-tailed and held to a significance level of alpha = 0.05. Post-hoc analyses will otherwise be conducted as appropriate pending the outcome of the initial primary analyses.
Change in anxiety, measured using the Generalized Anxiety Disorder-7 | Baseline to up to 10 weeks
  Skewed data will be log transformed or other appropriate transformations performed as necessary. Simple associations between demographic variables and outcome variables will be conducted to determine the need for control variables. Significant pre- to post-intervention change in psychosocial outcomes will be analyzed using the repeated measures linear mixed model. All analyses will be two-tailed and held to a significance level of alpha = 0.05. Post-hoc analyses will otherwise be conducted as appropriate pending the outcome of the initial primary analyses.
Change in coping style, assessed using the Brief Cope scale | Baseline to up to 10 weeks
  Skewed data will be log transformed or other appropriate transformations performed as necessary. Simple associations between demographic variables and outcome variables will be conducted to determine the need for control variables. Significant pre- to post-intervention change in psychosocial outcomes will be analyzed using the repeated measures linear mixed model. All analyses will be two-tailed and held to a significance level of alpha = 0.05. Post-hoc analyses will otherwise be conducted as appropriate pending the outcome of the initial primary analyses.
Change in depression assessed using the Patient Health Questionnaire depression module-9 | Baseline to up to 10 weeks
  Skewed data will be log transformed or other appropriate transformations performed as necessary. Simple associations between demographic variables and outcome variables will be conducted to determine the need for control variables. Significant pre- to post-intervention change in psychosocial outcomes will be analyzed using the repeated measures linear mixed model. All analyses will be two-tailed and held to a significance level of alpha = 0.05. Post-hoc analyses will otherwise be conducted as appropriate pending the outcome of the initial primary analyses.
Change in distress assessed using the Distress Thermometer measure | Baseline to up to 10 weeks
  Skewed data will be log transformed or other appropriate transformations performed as necessary. Simple associations between demographic variables and outcome variables will be conducted to determine the need for control variables. Significant pre- to post-intervention change in psychosocial outcomes will be analyzed using the repeated measures linear mixed model. All analyses will be two-tailed and held to a significance level of alpha = 0.05. Post-hoc analyses will otherwise be conducted as appropriate pending the outcome of the initial primary analyses.
Change in fatigue assessed using the FACIT | Baseline to up to 10 weeks
  Skewed data will be log transformed or other appropriate transformations performed as necessary. Simple associations between demographic variables and outcome variables will be conducted to determine the need for control variables. Significant pre- to post-intervention change in psychosocial outcomes will be analyzed using the repeated measures linear mixed model. All analyses will be two-tailed and held to a significance level of alpha = 0.05. Post-hoc analyses will otherwise be conducted as appropriate pending the outcome of the initial primary analyses.
Change in Hispanic-specific stress measured using the abbreviated version of the Hispanic Stress Inventory-Immigrant version | Baseline to up to 10 weeks
  Skewed data will be log transformed or other appropriate transformations performed as necessary. Simple associations between demographic variables and outcome variables will be conducted to determine the need for control variables. Significant pre- to post-intervention change in psychosocial outcomes will be analyzed using the repeated measures linear mixed model. All analyses will be two-tailed and held to a significance level of alpha = 0.05. Post-hoc analyses will otherwise be conducted as appropriate pending the outcome of the initial primary analyses.
Change in perceived stress measured using the Perceived Stress Scale | Baseline to up to 10 weeks
  Skewed data will be log transformed or other appropriate transformations performed as necessary. Simple associations between demographic variables and outcome variables will be conducted to determine the need for control variables. Significant pre- to post-intervention change in psychosocial outcomes will be analyzed using the repeated measures linear mixed model. All analyses will be two-tailed and held to a significance level of alpha = 0.05. Post-hoc analyses will otherwise be conducted as appropriate pending the outcome of the initial primary analyses.
Change in quality of life as measured using the Functional Assessment Chronic Illness Therapy (FACIT)-General | Baseline to up to 10 weeks
  Skewed data will be log transformed or other appropriate transformations performed as necessary. Simple associations between demographic variables and outcome variables will be conducted to determine the need for control variables. Significant pre- to post-intervention change in psychosocial outcomes will be analyzed using the repeated measures linear mixed model. All analyses will be two-tailed and held to a significance level of alpha = 0.05. Post-hoc analyses will otherwise be conducted as appropriate pending the outcome of the initial primary analyses.
Change in self-efficacy measured using the Spanish Chronic Disease Self-Efficacy scale | Baseline to up to 10 weeks
  Skewed data will be log transformed or other appropriate transformations performed as necessary. Simple associations between demographic variables and outcome variables will be conducted to determine the need for control variables. Significant pre- to post-intervention change in psychosocial outcomes will be analyzed using the repeated measures linear mixed model. All analyses will be two-tailed and held to a significance level of alpha = 0.05. Post-hoc analyses will otherwise be conducted as appropriate pending the outcome of the initial primary analyses.
Change in social support assessed using the Medical Outcomes Study-Social Support Survey | Baseline to up to 10 weeks
  Skewed data will be log transformed or other appropriate transformations performed as necessary. Simple associations between demographic variables and outcome variables will be conducted to determine the need for control variables. Significant pre- to post-intervention change in psychosocial outcomes will be analyzed using the repeated measures linear mixed model. All analyses will be two-tailed and held to a significance level of alpha = 0.05. Post-hoc analyses will otherwise be conducted as appropriate pending the outcome of the initial primary analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Ceballos, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States